CLINICAL TRIAL: NCT04344366
Title: Association Between Early Childhood Caries, Low Birth Weight and Nutritional Risk Factors: (Cohort Study)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, dina farrag morad, principle investigator, Cairo University
Other Study IDs: ECC in LBW children
Record Dates: First submitted 2020-02-05; First posted 2020-04-14 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: ECC; LBW Children
Keywords: ECC; premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: children with low birth weight
- group B: children with normal birth weight

SUMMARY:
The aim of this study is to assess the ECC experience in children aged from 12 to 36 month with low birth weight children in comparison to normal birth weight.

DETAILED DESCRIPTION:
Dental caries is on the top list of most widespread chronic diseases in addition to be a major public health issue. Dental caries is the single most common chronic childhood disease; it is 5 times more common than asthma, 7 times more common than hay fever and 14 times more common than chronic bronchitis. Deciduous tooth decay was ranked as the 12th most prevalent condition, affecting 560 million children in the 2015 Global Burden of Disease Study.

Low birth weight and premature birth are highly related to infant mortality, perinatal infections and the poor growth and development of children. Some risk groups have been identified, and attention should be focused on them so that preventive and health promotion measures are taken in an attempt to reverse this situation. One of these risk groups is composed of children born prematurely. Prematurity may be a predisposing factor for the development of caries.

There is a strong relationship between birth weight and infant mortality and morbidity and chronic diseases later in life. Many studies discussed the association between birth weight and dental caries however the results were conflicting. Knowledge of the association between low birth weight and the risk factors of ECC and the associated nutritional risk factors will improve the preventive and health promotion measures for this population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children.
* Children aged from 12 to 36 month.

Exclusion Criteria:

* Refusal of participation from the parents.
* Medically compromised children
* Major illness
* Child with special needs
* Any systemic disease that may affect caries experience.
* Any congenital deformity that may affect caries experience.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy, children aged from 12 to 36 month.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
early childhood caries | 1 year
  Dental examination

SECONDARY OUTCOMES:
Nutritional risk factors | 1 year
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ola Omar, Study Director — Professor of Pediatric Dentistry and Dental Public Health; Marwa Ali, Study Chair — Lecturer of Pediatric Dentistry and Dental Public Health

REFERENCES:
- [Background] da Silva Castro CR, de Sousa Cabral MBB, Mota ELA, Cangussu MCT, Vianna MIP. Analysis of the influence of low birth weight on the time of eruption of dental caries in children in early childhood. J Public Health Dent. 2019 Dec;79(4):292-297. doi: 10.1111/jphd.12322. Epub 2019 May 13. PMID 31087372
- [Background] Masumo R, Birungi N, Bardsen A, Fadnes LT, Astrom AN. Impact of low birthweight on early childhood caries in 6-36 months old infants in Uganda: A cross-sectional study. Acta Odontol Scand. 2014 May;72(4):312-20. doi: 10.3109/00016357.2014.880189. Epub 2014 Jan 27. PMID 24460034